CLINICAL TRIAL: NCT05205317
Title: Comparison of the Therapeutic Effects of Vaginal Repair and Vaginal Repair + Metformin in the Treatment of Cesarean Section Scar Defect
Brief Title: Comparison of the Therapeutic Effects of VR and VR + Metformin in the Treatment of Cesarean Section Scar Defect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-21-012
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Defect
Keywords: cesarean section scar defect; metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaginal repair + metformin (Experimental): CSD patients were treated with vaginal repair of CSD in combination with metformin (Boke, 500 mg, Wanhui Shuanghe, Beijing, China) as an oral medicine (abbreviated as VR + metformin). In the group of VR + metformin, the patients start oral metformin from one month before the operation to 6 months after the operation. The dose is 500mg twice a day. The detailed procedure of VR has been described in investigators' previous study.
  Interventions: Drug: Metformin Hydrochloride Sustained-release Tablets; Procedure: Vaginal repair
- vaginal repair (Active Comparator): The procedure of vaginal repair of CSD was shown as following. The bladder was dissected away carefully from the uterus toward the abdominal cavity until the peritoneum was reached. The CSD tissue was cut to the normal healthy muscle after the abdominal cavity had been entered, and the lower uterine segments had been completely exposed. A double layer of 1-0 absorbable interrupted sutures was used to close the incisions.
  Interventions: Procedure: Vaginal repair

INTERVENTIONS:
Drug: Metformin Hydrochloride Sustained-release Tablets — drug
  Other Names: Boke
  Arms: vaginal repair + metformin
Procedure: Vaginal repair — The procedure of vaginal repair of CSD was shown as following. The bladder was dissected away carefully from the uterus toward the abdominal cavity until the peritoneum was reached. The CSD tissue was cut to the normal healthy muscle after the abdominal cavity had been entered, and the lower uterine segments had been completely exposed. A double layer of 1-0 absorbable interrupted sutures was used to close the incisions.

SUMMARY:
Cesarean section scar defect (CSD) is a novel recognized cause of postmenstrual abnormal uterine bleeding in women. No clinical guidelines have been issued for the management of CSD. The investigators have previously demonstrated that vaginal repair of CSD was an relative effective treatment of CSD. However, only 28.2% of the CSD patients normalized to less than 7 days of menstruation, whereas 51.2% of women had 7 to 10 days of menstruation at 6 months post vaginal repair. The previous research suggested that the occurrence of CSD may be related to the aging phenotype of the myometrium. Metformin, as a classic diabetes treatment drug, has an important position in anti-aging therapy. Therefore, the randomized study was designed to evaluate whether the application of metformin in combination with vaginal repair could achieve better clinical effects than those achieved by vaginal CSD repair alone.

DETAILED DESCRIPTION:
The previous research suggested that the occurrence of cesarean section scar defect (CSD) may be related to the aging phenotype of the myometrium. The aging of the myometrium in some cesarean section patients reduces the proliferation and repair of smooth muscle cells and endometrial cells to a certain extent. The prognosis of vaginal repair is poor and the repair of the endometrium during menstruation is not good.

Metformin, as a classic diabetes treatment drug, has an important position in anti-aging therapy. Its research and application range is the widest, and significant results have been achieved in a number of clinical trials. At the same time, its side effects are less than other anti-aging drugs, and the patient adaptability is better. It maybe the best choice for the treatment of anti-aging diseases. Therefore, the randomized study was designed to evaluate whether the application of metformin in combination with vaginal repair could achieve better clinical effects than those achieved by vaginal CSD repair alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are younger than 40 and over the age of 18.
2. Clearly diagnosed with CSD.
3. Experiencing clinical features of abnormal uterine bleeding, prolonged menstrual flow (the duration of menstruation is more than 10 days).
4. The thickness of the remaining muscular layer of CSD was less than 3 mm.
5. Normal range of blood sugar and insulin
6. No serious medical problems (important viscera function in the normal range).
7. No uterine fibroids, endometriosis, adenomyosis
8. No malignant tumors.
9. Sign the informed consent.

Exclusion Criteria:

1. Over the age of 40 or younger than 18;
2. Indefinite diagnosis.
3. Malignant tumors.
4. With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
5. Contraindications to metformin (baseline creatinine >124μmol/L, hypersensitivity to metformin, or a metabolic acidosis), use of drugs that might interact with metformin (glyburide, furosemide, or cationic drugs)
6. Pregnant.
7. Mental diseases.
8. Unwilling to comply with the research plan.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of menstruation (day) | 6 months after vaginal repair of CSD
  Duration of menstruation (day)
thickness of the remaining muscular layer (TRM) (mm) | 6 months after vaginal repair of CSD
  The thickness of the remaining muscular layer is measured by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Subsequent pregnancy outcomes | At least 1 year after vaginal repair of CSD
  Subsequent pregnancy outcomes
Duration of menstruation (day) | At least 1 year after vaginal repair of CSD
  Duration of menstruation (day)

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No